CLINICAL TRIAL: NCT02919111
Title: Gallium-68 PSMA-11 PET in Intermediate to High-risk Preprostatectomy Patients
Acronym: PSMA PreRP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Thomas Hope, Assistant Professor of Radiology and Biomedical Imaging, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16559; NCI-2018-00038 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2016-09-26; First posted 2016-09-29 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ga-68 labeled PSMA-11 PET (Experimental): PSMA PET imaging: Patients will receive Ga-68 labeled PSMA-11 PET and then undergo PET/CT or PET/MRI approximately 55-70 minutes later.
  Interventions: Drug: Ga-68 labeled PSMA-11 PET

INTERVENTIONS:
Drug: Ga-68 labeled PSMA-11 PET — Patients will be imaged using Ga-68 labeled PSMA-11 PET to determine if the presence of metastatic disease. Prostate Specific Membrane Antigen (PSMA) is a protein expressed on prostate cancer cells that can be imaged using small molecules that target this protocol.
  Other Names: Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled Glu-NH-CO-NH- Lys(Ahx)-HBED-CC; Ga-68 labeled Glu-urea- Lys(Ahx)-HBED-CC; Ga-68 labeled HBED-CC PSMA

SUMMARY:
The investigators are imaging patients with prostate cancer using a new PET imaging agent (Ga-68-PSMA-11) in order to evaluate it's ability to detection prostate cancer in patients with high risk disease prior to prostatectomy.

DETAILED DESCRIPTION:
Imaging and staging of prostate cancer is critical for surgical and treatment planning. Patients with suspected metastatic prostate cancer will be imaged using Gallium-68 labeled PSMA-11 in order to demonstrate its utility. The investigators plan to utilize this data to obtain further approvals of the Ga-68-PSMA-11 compound, so that this agent will become available for clinical imaging in prostate cancer patients. In the pre-prostatectomy population, the primary objective is to determine the sensitivity and specificity for detection on nodal metastasis.

This compound has been shown to be superior to choline based PET agents for the staging of prostate cancer, both Carbon-11 and Fluorine-18 compounds. But this compound was not patented and therefore no company or private entity will make the investment required to bring Ga-68-PSMA-11 to market. In the vacuum of availability, academic groups must take the lead in order to collect the necessary data for future FDA approval.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate adenocarcinoma.
* Planned prostatectomy with lymph node dissection.
* Intermediate to high-risk disease (as determined by elevated Prostate-specific antigen (PSA) [PSA>10], T-stage [T2b or greater], Gleason score [Gleason score > 6] or other risk factors).
* Diagnostic CT or MRI as part of the PET study or performed within one month of PSMA PET.
* Karnofsky performance status of greater than 50 (or Eastern Cooperative Oncology Group (ECOG) /World Health Organization (WHO) equivalent).
* Age > 18.
* Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

* Patients not capable of getting PET study due to weight, claustrophobia, or inability to lay still for the duration of the exam.
* Neoadjuvant chemotherapy or radiation therapy prior to prostatectomy.
* Including focal ablation techniques (HiFu).
* Androgen deprivation therapy or other neoadjuvant treatments prior to PET imaging and surgery.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Djaileb L, Armstrong WR, Thompson D, Gafita A, Farolfi A, Rajagopal A, Grogan TR, Nguyen K, Benz MR, Hotta M, Barbato F, Ceci F, Schwarzenbock SM, Unterrainer M, Zacho HD, Juarez R, Cooperberg M, Carroll P, Washington S, Reiter RE, Eiber M, Herrmann K, Fendler WP, Czernin J, Hope TA, Calais J. Presurgical 68Ga-PSMA-11 Positron Emission Tomography for Biochemical Recurrence Risk Assessment: A Follow-up Analysis of a Multicenter Prospective Phase 3 Imaging Trial. Eur Urol. 2023 Dec;84(6):588-596. doi: 10.1016/j.eururo.2023.06.022. Epub 2023 Jul 21. PMID 37482512
- [Derived] Hope TA, Eiber M, Armstrong WR, Juarez R, Murthy V, Lawhn-Heath C, Behr SC, Zhang L, Barbato F, Ceci F, Farolfi A, Schwarzenbock SM, Unterrainer M, Zacho HD, Nguyen HG, Cooperberg MR, Carroll PR, Reiter RE, Holden S, Herrmann K, Zhu S, Fendler WP, Czernin J, Calais J. Diagnostic Accuracy of 68Ga-PSMA-11 PET for Pelvic Nodal Metastasis Detection Prior to Radical Prostatectomy and Pelvic Lymph Node Dissection: A Multicenter Prospective Phase 3 Imaging Trial. JAMA Oncol. 2021 Nov 1;7(11):1635-1642. doi: 10.1001/jamaoncol.2021.3771. PMID 34529005

RESULTS

PARTICIPANT FLOW:
Groups:
- Ga-68 Labeled PSMA-11 PET: PSMA Positron Emission Tomography (PET) imaging: Patients will receive Ga-68 labeled PSMA-11 PET and then undergo PET/CT or PET/MRI approximately 55-70 minutes later.
  Ga-68 labeled PSMA-11 PET: Patients will be imaged using Ga-68 labeled PSMA-11 PET to determine if the presence of metastatic disease. Prostate Specific Membrane Antigen (PSMA) is a protein expressed on prostate cancer cells that can be imaged using small molecules that target this protocol.
Period: Overall Study
Arm/Group | Ga-68 Labeled PSMA-11 PET
Started | 299
Completed | 299
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 299
Age, Customized [Count of Participants; unit: Participants]
  40-49 years old | 3
  50-59 years old | 25
  60-69 years old | 126
  70-79 years old | 124
  80-89 years old | 19
  90-99 years old | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 299
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 262
  Unknown or Not Reported | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 19
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 8
  White | 218
  More than one race | 1
  Unknown or Not Reported | 47
Region of Enrollment [Number; unit: participants]
  United States | 299

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of PSMA PET for the Detection of Regional Nodal Metastases Compared to Pathology at Radical Prostatectomy
Description: Sensitivity is defined as the ratio of the proportion of the patients who have the condition of interest and whose test results are positive over the number who have the disease. Patients who have a positive node on imaging and on pathology will be considered a true-positive. Patients who have no nodes on imaging and pathology will be considered true-negatives. Patients with positive nodes on imaging and negative on pathology will be considered false positives and those with positive nodes on pathology but negative on imaging will be considered false negatives. Follow-up scans for up to one year can be used in analysis
Time Frame: Up to 1 year
Measure: Number; unit: proportion of participants
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 299
proportion of participants | .43

2. Primary Outcome: Specificity of of PSMA PET for the Detection of Regional Nodal Metastases Compared to Pathology at Radical Prostatectomy
Description: Specificity is defined as the number of non-diseased participants correctly classified divided by all non-diseased individuals. Patients who have a positive node on imaging and on pathology will be considered a true-positive. Patients who have no nodes on imaging and pathology will be considered true-negatives. Patients with positive nodes on imaging and negative on pathology will be considered false positives and those with positive nodes on pathology but negative on imaging will be considered false negatives. Follow-up scans for up to one year can be used in analysis
Time Frame: Up to 1 year
Measure: Number; unit: proportion of participants
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 299
proportion of participants | .94

3. Primary Outcome: Positive Predictive Value (PPV) of of PSMA PET for the Detection of Regional Nodal Metastases Compared to Pathology at Radical Prostatectomy
Description: PPV is the proportion of patients with positive test who actually have the disease. Patients who have a positive node on imaging and on pathology will be considered a true-positive. Patients who have no nodes on imaging and pathology will be considered true-negatives. Patients with positive nodes on imaging and negative on pathology will be considered false positives and those with positive nodes on pathology but negative on imaging will be considered false negatives. Follow-up scans for up to one year can be used in analysis
Time Frame: Up to 1 year
Measure: Number; unit: proportion of true positives
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 299
proportion of true positives | .64

4. Primary Outcome: Negative Predictive Value (NPV) of PSMA PET for the Detection of Regional Nodal Metastases Compared to Pathology at Radical Prostatectomy
Description: NPV is the ratio of participants truly diagnosed as negative to all those who had negative test results. Patients who have a positive node on imaging and on pathology will be considered a true-positive. Patients who have no nodes on imaging and pathology will be considered true- negatives. Patients with positive nodes on imaging and negative on pathology will be considered false positives and those with positive nodes on pathology but negative on imaging will be considered false negatives. Follow-up scans for obtained up to one year after study scan be used in analysis.
Time Frame: Up to 1 year
Measure: Number; unit: proportion of true negatives
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 299
proportion of true negatives | .87

5. Secondary Outcome: Number of Participants With Grade 3 Treatment-related Adverse Events
Description: All grade 3 and above adverse events were recorded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0. The Investigator assigns grade, attribution of the possible association of the event with use of the investigational drug. The safety parameters include spontaneous reports of adverse events reported to the investigator by patients
Time Frame: Up to 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 299
Participants | 0

6. Secondary Outcome: Sensitivity of PSMA PET for the Detection of Extra-pelvic Nodal Metastases
Description: Gallium 68 labeled PSMA-11 (68Ga-PSMA-11) positive lymph nodes will be considered for detection of extra-pelvic nodal metastases and assessed by change in size. Participants who if on follow-up imaging within 3-12 months, have lymph nodes which decrease by more than 30% or increase by more than 20% in short axis diameter (with a minimum of 3 mm in change in size) or with solitary lymph node regions show a decrease of Prostate-specific antigen (PSA) by >50% after targeted treatment and the lymph nodes do not change in size (less than 30% decrease or less than 20% increase in short axis diameter) will be counted as true positives. If on follow-up imaging, sites of initial 68Ga-PSMA-11 positive lymph node lesions < 30% without systemic therapy or focal therapy at this site or if 68Ga-PSMA-11 positive lymph node lesions that do not meet criteria for above false positive or true positive will be counted as false positives.
Time Frame: Up to 1 year
Population: Data on the detection of extra-pelvic nodal metastases was not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

7. Secondary Outcome: Specificity of PSMA PET for the Detection of Extra-pelvic Nodal Metastases
Description: 68Ga-PSMA-11 positive lymph nodes will be considered for detection of extra-pelvic nodal metastases and assessed by change in size. Participants who if on follow-up imaging within 3-12 months, have lymph nodes which decrease by more than 30% or increase by more than 20% in short axis diameter (with a minimum of 3 mm in change in size) or with solitary lymph node regions show a decrease of PSA by >50% after targeted treatment and the lymph nodes do not change in size (less than 30% decrease or less than 20% increase in short axis diameter) will be counted as true positives. If on follow-up imaging, sites of initial 68Ga-PSMA-11 positive lymph node lesions < 30% without systemic therapy or focal therapy at this site or if 68Ga-PSMA-11 positive lymph node lesions that do not meet criteria for above false positive or true positive will be counted as false positives.
Time Frame: Up to 1 year
Population: Data on the detection of extra-pelvic nodal metastases was not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

8. Secondary Outcome: Positive Predictive Value of PSMA PET for the Detection of Extra-pelvic Nodal Metastases
Description: as for outcome 7
Time Frame: Up to 1 year
Population: Data on the detection of extra-pelvic nodal metastases was not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

9. Secondary Outcome: Negative Predictive Value of PSMA PET for the Detection of Extra-pelvic Nodal Metastases
Description: as for outcome 7
Time Frame: Up to 1 year
Population: Data on the detection of extra-pelvic nodal metastases was not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

10. Secondary Outcome: Sensitivity of PSMA PET for the Detection of Visceral Metastases
Description: Visceral lesions (non-lymph node soft tissue or organ) will be assessed by change in size. 68Ga-PSMA-11 positive visceral lesions will be considered True positive if on follow-up imaging within 3-12 months, visceral lesions seen on imaging decrease by 30% (for patients undergoing systemic treatment of focal therapy at this site) or increase by 20% in largest diameter or if participants with solitary visceral metastasis show a decrease of PSA by greater than 50% after targeted treatment and lesions do not change in size (less than 30% decrease or 20% increase in largest diameter) and False positive if on follow-up imaging within 3-12 months, sites of initial 68Ga-PSMA-11 positive visceral lesions seen on CT or MRI decrease by more than 30% without systemic therapy or focal therapy at this site or if 68Ga-PSMA-11 positive visceral lesions do not meet the criteria for above false positive or true positive findings.
Time Frame: Up to 1 year
Population: Data on the detection of visceral metastases was not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

11. Secondary Outcome: Specificity of PSMA PET for the Detection of Visceral Metastases
Description: as for outcome 10
Time Frame: Up to 1 year
Population: Data on the detection of visceral metastases was not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

12. Secondary Outcome: Positive Predictive Value of PSMA PET Visceral Metastases
Description: as for outcome 10
Time Frame: Up to 1 year
Population: Data on the detection of visceral metastases was not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

13. Secondary Outcome: Negative Predictive Value of PSMA PET for the Detection of Visceral Metastases
Description: as for outcome 10
Time Frame: Up to 1 year
Population: Data on the detection of visceral metastases was not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

14. Secondary Outcome: Sensitivity of PSMA PET for the Detection of Osseous Metastases
Description: 68Ga-PSMA-11 positive bone lesions will be considered a True positive if there was a corresponding positive sclerotic lesion on the CT portion of the 68Ga-PSMA-11 PET in the same location as the PSMA uptake, If there is focal uptake seen in the same location as the PSMA uptake on the baseline bone scan performed within one month of 68Ga-PSMA-11 PET, if there is a lesion noted in the same location as the PSMA uptake on the initial MRI performed within one month of 68Ga-PSMA-11 PET, if within 12 months follow-up CT demonstrates development of sclerosis in the same location as the PSMA uptake, if within 12 months follow-up MRI demonstrates a new bone lesion in the same location as the PSMA uptake, if within 12 months follow-up bone scan demonstrates new focal uptake in the same location as the PSMA uptake and a False positive if 68Ga-PSMA-11 positive bone lesions do not meet the criteria for true positive findings.
Time Frame: Up to 1 year
Population: Data on the detection of osseous metastases was not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

15. Secondary Outcome: Specificity of PSMA PET for the Detection of Osseous Metastases
Description: as for outcome 14
Time Frame: Up to 1 year
Population: Data on the detection of osseous metastases was not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

16. Secondary Outcome: Positive Predictive Value of PSMA PET for the Detection of Osseous Metastases
Description: as for outcome 14
Time Frame: Up to 1 year
Population: Data on the detection of osseous metastases was not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

17. Secondary Outcome: Negative Predictive Value of PSMA PET for the Detection of Osseous Metastases
Description: as for outcome 14
Time Frame: Up to 1 year
Population: Data on the detection of osseous metastases was not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 3 days
Description: All grade 3 and above adverse events were reported
Arm/Group | Ga-68 Labeled PSMA-11 PET
All-Cause Mortality (participants affected / at risk) | 0/299
Serious Adverse Events (participants affected / at risk) | 0/299
Other Adverse Events (participants affected / at risk) | 0/299

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT02919111/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT02919111/ICF_001.pdf